CLINICAL TRIAL: NCT05157035
Title: Testing a Mindfulness/Acceptance-Based Smartphone App Intervention to Develop Resilience Among Nurses Traumatized From the Effects of the COVID-19 Pandemic: A Randomized Controlled Trial
Brief Title: Testing a Mindfulness/Acceptance-Based Smartphone App for Nurses Impacted by the COVID-19 Pandemic
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Andrew Thomas Reyes, Assistant Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1760618-3
Record Dates: First submitted 2021-12-09; First posted 2021-12-14 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Posttraumatic Stress Disorder
Keywords: posttraumatic stress disorder; mindfulness; COVID-19; mindfulness app
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; COVID-19 | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Mindfulness/Acceptance-Based Smartphone App (MABSA) Intervention Group will use the smartphone app which comprises of audio-guided mindfulness meditations and video lessons. Participants are asked to listen to at least one guided meditation daily and watch one video lesson each week. Participants will also receive a weekly phone call for emotional and technical support. The wait-list control group will have the option to use the app-based intervention after 10 weeks of being in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness/Acceptance-Based Smartphone App (MABSA) Intervention Group (Experimental): The intervention is 6 weeks in duration. Participants will be asked to listen daily to at least one audio-guided mindfulness meditation embedded in the app. They will also be asked to watch a weekly video lesson on mindfulness and acceptance and will be asked to write a reflection about the video. They will also receive weekly emotional and technical support during the duration of the intervention.
  Interventions: Behavioral: Mindfulness/Acceptance-Based Smartphone App (MABSA)
- Wait-List Control Group (No Intervention): The control group is a wait-list control group. Participants in the control group will be offered to use the app after 10 weeks of being in the study. The control group participants once they opted to use the app after 10 weeks will only have access to the app for 6 weeks.

INTERVENTIONS:
Behavioral: Mindfulness/Acceptance-Based Smartphone App (MABSA) — This is a mindfulness- and acceptance-based smartphone app. The mindfulness and acceptance exercises embedded in the app are based on the principles of Acceptance and Commitment Therapy. Participants in the intervention group will be using the app for 6 weeks. They are expected to access the meditations and mindfulness exercises within the app on a daily basis.
  Arms: Mindfulness/Acceptance-Based Smartphone App (MABSA) Intervention Group

SUMMARY:
The purpose of the study is to test the feasibility and acceptability of a mindfulness- and acceptance-based smartphone app (MABSA) intervention for frontline nurses emotionally and psychologically impacted by the COVID-19 pandemic. The study will use a randomized controlled trial design of two groups: an intervention group of about 30 participants with posttraumatic stress symptoms and a wait-list control group of about 30 participants. The duration of the MABSA intervention is 6 weeks. The following are the outcomes to be measured: resilience, PTSD, mindfulness, experiential avoidance, and rumination.

DETAILED DESCRIPTION:
The objective of the proposed study is to evaluate the feasibility of the Mindfulness/Acceptance-Based Smartphone App (MABSA) intervention in a randomized controlled trial (RCT) environment and to obtain generalized information (i.e., initial efficacy, recruitment, retention, adherence, satisfaction, and usability of the refined intervention). The expected results will provide the foundation for a prospective, fully powered, larger-scale RCT study. The investigator previously developed the MABSA and pilot-tested it in a single-arm study among veterans, and the study will be testing the app among nurses who have been emotionally and psychologically impacted by the COVID-19 pandemic. Our central hypothesis is that the refined MABSA intervention would improve intervention satisfaction, app usability, and adherence and positively affect resilience, PTSD, mindfulness, experiential avoidance, and rumination. The specific aims of the proposed study are outlined below.

AIM 1: To refine the previously developed MABSA intervention. The 6-week smartphone-delivered program will involve (1) daily audio-guided meditations on various mindfulness and acceptance exercises constructed based on the principles of acceptance and commitment therapy; (2) weekly support and feedback through phone calls and/or texting the intervention facilitators; and (3) ecological momentary assessment (daily monitoring of PTSD and resilience) to monitor the progression of treatment response (i.e., the trajectory of resilience and PTSD recovery). The investigator will obtain qualitative feedback on program content and format through a pilot test of the prototype with a group of eligible nurses (N = 4). Upon revising the intervention based on participants' feedback, the investigator will develop the intervention protocol manual for the RCT.

AIM 2: To test the feasibility and acceptability of the refined MABSA intervention in a small-scale RCT for a prospective, fully powered, larger-scale RCT study. The small-scale RCT study will involve the following two groups of frontline nurses: (1) the MABSA intervention group (N = 30) and the wait-list control group (N = 30). Upon collecting the data on recruitment, retention, adherence, intervention satisfaction, and app usability, the study will determine the preliminary efficacy based on the following five outcomes: resilience, PTSD, mindfulness, experiential avoidance, and rumination. Qualitative feedback on the facilitators of and challenges to recruitment, retention, and adherence will be collected via exit interviews.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged 18 years old or older, (2) frontline registered nurse or licensed practical nurse practising in the United States, (3) has at least daily access to their own Apple iPhone (version 5 or later) or Android phone, and (4) have posttraumatic stress disorder (PTSD) symptoms (must have a score of 33 or above on the PTSD Checklist for DSM-5)

Exclusion Criteria:

* (1) Those who have a score of 32 or below on the PTSD Checklist for DSM-5, and (2) healthcare workers that are not RNs or LPNs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-10-14 (Estimated); Study Completion 2022-10-14 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Symptoms (PTSD Checklist for DSM-5 or also called PCL-20) | The investigator will measure PTSD at baseline, mid-intervention (Week 3), post-intervention (Week 6), and at one-month follow-up
  Changes in posttraumatic stress disorder (PTSD) symptoms based on the PTSD Checklist for DSM-5 (PCL-20). There are 20 items in the PCL-20. The minimum value of PCL-20 is 0, and the maximum value is 80. Higher scores mean a worse outcome (more severe symptoms of Posttraumatic Stress Disorder).
Resilience (Connor-Davidson Resilience Scale or also called CD-RISC-25) | The investigator will measure resilience (Connor-Davidson Resilience Scale, CD-RISC-25) at baseline, mid-intervention (Week 3), post-intervention (Week 6), and at one-month follow-up
  Changes in resilience based on the Connor-Davidson Resilience Scale (CD-RISC-25). There are 25 items in the CD-RISC-25. The minimum value of CD-RISC-25 is 0, and the maximum value is 100. Higher scores mean a better outcome (higher level of resilience).
Mindfulness (Mindfulness Attention and Awareness Scale or also called MAAS) | The investigator will measure mindfulness (Mindfulness Attention and Awareness Scale, MAAS) at baseline, mid-intervention (Week 3), post-intervention (Week 6), and at one-month follow-up
  Changes in mindfulness based on the Mindfulness Attention and Awareness Scale (MAAS). There are 15 items in the MAAS. The minimum value of MAAS is 15, and the maximum value is 90. Higher scores mean a better outcome (higher level of mindfulness).
Experiential Avoidance (Acceptance and Action Questionnaire or also called AAQ) | The investigator will measure experiential avoidance (Acceptance and Action Questionnaire, AAQ) at baseline, mid-intervention (Week 3), post-intervention (Week 6), and at one-month follow-up
  Changes in experiential avoidance based on the Acceptance and Action Questionnaire (AAQ). There are 7 items in the AAQ. The minimum value of the AAQ is 7, and the maximum value is 49. Higher scores mean a worse outcome (higher level of experiential avoidance or the unwillingness to be present with difficult emotions and thoughts).
Rumination (Rumination Response Scale or also called RRS) | The investigator will measure rumination (Rumination Response Scale, RRS) at baseline, mid-intervention (Week 3), post-intervention (Week 6), and at one-month follow-up
  Changes in rumination based on the Rumination Response Scale (RRS). The RRS has 22 items. The minimum value of the RRS is 22, and the maximum value is 88. Higher scores mean a worse outcome (higher level of rumination or perseverative and passive focus on symptoms and the possible causes and outcomes of psychological distress)

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Recovery (Abbreviated Version of the Posttraumatic Stress Disorder Checklist or also called PCL-8) | The investigator will measure posttraumatic stress disorder symptoms daily using the app (ecological momentary assessment).
  Daily measures of posttraumatic stress disorder (PTSD) using the abbreviated PTSD Checklist for DSM-5 (PCL-8). The PCL-8 is a shortened version of the PCL-20. There are 8 items in the PCL-8. The minimum value is 0, and the maximum value is 32. Higher scores mean a worse outcome (greater severity of Posttraumatic Stress Disorder symptoms).
Resilience Progression (Abbreviated Version of the Connor-Davidson Resilience Scale or also called CD-RISC-10) | The investigator will measure resilience daily using the app (ecological momentary assessment)
  Daily measures of resilience using the abbreviate Connor-Davidson Resilience Scale 10 (CD-RISC-10). There are 10 items in the CD-RISC-10. The minimum value of the CD-RISC-10 is 0, and the maximum value is 40. Higher scores mean a better outcome (higher level of resilience).

OTHER OUTCOMES:
Intervention Satisfaction (Intervention Satisfaction Survey or also called ISS). | The investigator will measure intervention satisfaction at mid-intervention (Week 3) and post-intervention (Week 6)
  The Intervention Satisfaction Survey (ISS) will be used to determine the degree of acceptability of the intervention (e.g., overall satisfaction, perceived helpfulness, comprehension, intentions to use, and perceived fit). There are 8 items in the ISS. The minimum value for the ISS is 8, and the maximum value is 48. Higher scores mean a better outcomes (indicating higher level of satisfaction with the app).
Usability of the App (System Usability Scale or also called SUS) | The investigator will measure perceived usability of the app at mid-intervention (Week 3) and post-intervention (Week 6)
  The perceived usability of the app will be measured using the System Usability Scale (SUS). There are 10 items in the SUS. The minimum value of the SUS is 10, and the maximum value is 50. Higher scores mean a better outcome (i.e., that the app is perceived to be useful and relevant for the participants).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reyes AT. The Process of Learning Mindfulness and Acceptance through the Use of a Mobile App Based on Acceptance and Commitment Therapy: A Grounded Theory Analysis. Issues Ment Health Nurs. 2022 Jan;43(1):3-12. doi: 10.1080/01612840.2021.1953652. Epub 2021 Aug 4. PMID 34346278
- [Background] Reyes AT, Song H, Bhatta TR, Kearney CA. Exploring the relationships between resilience, mindfulness, and experiential avoidance after the use of a mindfulness- and acceptance-based mobile app for posttraumatic stress disorder. Perspect Psychiatr Care. 2022 Apr;58(2):776-784. doi: 10.1111/ppc.12848. Epub 2021 May 20. PMID 34018197
- [Background] Reyes AT. A Mindfulness Mobile App for Traumatized COVID-19 Healthcare Workers and Recovered Patients: A Response to "The Use of Digital Applications and COVID-19". Community Ment Health J. 2020 Oct;56(7):1204-1205. doi: 10.1007/s10597-020-00690-9. Epub 2020 Aug 9. No abstract available. PMID 32772205
- [Background] Reyes AT, Bhatta TR, Muthukumar V, Gangozo WJ. Testing the acceptability and initial efficacy of a smartphone-app mindfulness intervention for college student veterans with PTSD. Arch Psychiatr Nurs. 2020 Apr;34(2):58-66. doi: 10.1016/j.apnu.2020.02.004. Epub 2020 Feb 18. PMID 32248935